CLINICAL TRIAL: NCT07220473
Title: The Moody Longevity Trial: Tirzepatide to Slow Biological Aging
Brief Title: Tirzepatide to Slow Biological Aging
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25-0169
Record Dates: First submitted 2025-10-15; First posted 2025-10-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Aging; LONGEVITY 1
Keywords: DNA Methylation; Biological Clock Deceleration; GLP-1 Agonist
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Active Comparator): Participants will receive Tirzepatide 2.5 mg weekly for 24 weeks, followed by a 12-week off-drug follow-up.
  Interventions: Drug: Zepbound
- Placebo (No Intervention): Participants will be monitored for a total of 36 weeks without receiving medication.

INTERVENTIONS:
Drug: Zepbound — Auto injectors with a 2.5 mg dosage are given subcutaneously weekly.
  Other Names: Tirzepatide
  Arms: Tirzepatide

SUMMARY:
This pilot clinical study aims to investigate the potential effects of tirzepatide on biological aging in older adults. In this novel study, 90 adults aged 55-70 years with an indication for tirzepatide weight-loss therapy will be randomized to receive either tirzepatide 2.5 mg subcutaneously (SC) weekly or no drug for 24 weeks, followed by 12 weeks off the drug. Since tirzepatide is already recognized as a highly effective weight-loss agent in this population, the primary focus will not be on measuring weight loss. Instead, the study will document the effects of tirzepatide on markers of aging, physical function, and overall health.

DETAILED DESCRIPTION:
Primary Objective To estimate the potential effect of tirzepatide on biological aging using epigenetic age (based on established DNA methylation-based clocks), among people 55-70 years of age with an indication for tirzepatide weight loss therapy.

The principal investigator (PI) will measure DNA methylation-based aging clocks (DNAmAge, DNAm PhenoAge, DNAm GrimAge and DunedinPACE) before and after a 24-W course of tirzepatide. The primary analysis will determine whether tirzepatide treatment leads to a statistically significant change in biological age as indicated by these clocks. The PI will specifically assess epigenetic age acceleration (epigenetic age minus chronological age) and the pace of aging metric.

Secondary and Exploratory Objectives

Among people 55-70 years of age with an indication for tirzepatide weight loss therapy, the is aim to:

1. Estimate self-reported tolerability and acceptability of tirzepatide during the study period
2. Estimate changes in BMI and weight over 24 W of tirzepatide therapy, and in off-drug follow-up, between W 24 and 36
3. Estimate changes in physical function over 24 W of tirzepatide and, in off-drug follow-up, between W 24 and 36
4. Estimate changes in inflammatory, aging and neurocognitive biomarker profiles over 24 W of tirzepatide therapy, and in off-drug follow-up, between W 24 and 36
5. Estimate changes in other biological hallmarks/markers of aging
6. Explore relationships between the above outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-70 years
2. BMI ≥ 30 kg/m² or ≥ 27 kg/m² if also with ≥ 1 weight-related comorbidity
3. If taking anti-inflammatory or blood-pressure-/lipid-/glucose-lowering medications, no change in dose for ≥12 weeks prior to entry and no plans to dose escalate for the study duration
4. Willing and able to provide written informed consent and undergo all required study procedures

Exclusion Criteria:

1. BMI >35 kg/m²
2. Uncontrolled or end-stage, comorbid, cardiometabolic disease, in the opinion of the site investigator
3. Significant neurocognitive impairment, in the opinion of the site investigator
4. Current or planned use of medications for the treatment of obesity, or medications likely to cause significant changes in weight, during the study period (see prohibited medications, section 6.0)
5. Use of insulin
6. Plans to newly engage in formal, intensive physical activity or diet (such as ketogenic or very low carbohydrate) programs during the study period
7. Active eating disorder
8. Use of human growth hormone, tesamorelin, supraphysiologic testosterone or estradiol (stable doses for contraception, hypogonadism or other indications for exogenous sex steroid replacement therapy permitted) or anabolic steroids <12 W prior to entry, unless on a stable dose for >24 W prior to entry, or plans to start any of these medications while on study
9. Active, severe delayed gastric emptying
10. Prior bariatric surgery or major gastric surgery or plans for weight reduction surgery while on study
11. Known diabetic retinopathy
12. Personal or first-degree relative history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
13. Untreated, poorly controlled or previously undiagnosed thyroid disease
14. History of chronic pancreatitis
15. History of suicidal attempts or active suicidal ideation, in the opinion of the site investigator
16. Known allergy/sensitivity to GLP-1RA or GIPRA
17. Use or planned use of any immunomodulatory therapy or investigational therapy during the study period or use of an investigational therapy within 30 days of entry
18. Any other medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation.
19. Pregnancy, nursing or plans for either during the study period

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in DNA Methylation-Based Biological Age | Immediately before and after the study visit at Weeks 4, 12, and 24
  Change in biological age as measured by DNA methylation-based aging clocks (DNAmAge, DNAm PhenoAge, DNAm GrimAge, and DunedinPACE) following tirzepatide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blackwell, MD, FACP, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No